CLINICAL TRIAL: NCT00338832
Title: Adapting a Physical Activity Intervention for Schizophrenia
Brief Title: Effectiveness of a Lifestyle Intervention for Increasing Physical Activity in Adults With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Veterans Medical Research Foundation (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Laurie A. Lindamer, Research Scientist, Veterans Medical Research Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH071539 (NIH); R34MH071539 (NIH); DAHBR 96-BHB
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Schizophrenia
Keywords: Lifestyle Intervention; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive the Physically Ready for Invigorating Movement Every Day program
  Interventions: Behavioral: Physically Ready for Invigorating Movement Every Day (PRIME)
- 2 (Active Comparator): Participants will receive the Program for Activity, Leisure Skills, and Socialization
  Interventions: Behavioral: Program for Activity, Leisure Skills, and Socialization (PALSS)

INTERVENTIONS:
Behavioral: Physically Ready for Invigorating Movement Every Day (PRIME) — The PRIME program is a lifestyle intervention focused on increasing physical activity. The intervention is cognitive/behaviorally based, 24-weeks in length, and a lifestyle PA intervention known to be effective in the general population of adults. The program has been modified based on theory and empirical findings about this special subgroup. All participants will attend 90-minute sessions weekly for the first 16 weeks, then biweekly for the remaining 8 weeks. PRIME sessions will focus on learning about PA, setting PA-related goals, and assessing short- and long-term goals. Goals may include early-stage process-oriented goals, such as reading about PA benefits or finding a walking partner.
  Arms: 1
Behavioral: Program for Activity, Leisure Skills, and Socialization (PALSS) — PALSS sessions will focus on motivating participants to engage in leisure and social activity. Sessions will include interactive, structured activity that will be led by a therapist, as well as unstructured leisure activities, such as board games, cards, general socialization, and viewing a travel video. Social and communication skills will not be explicitly taught or practiced. All participants will attend 90-minute sessions weekly for the first 16 weeks, then biweekly for the remaining 8 weeks.
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of a lifestyle intervention in increasing physical activity and reducing disease symptoms in sedentary adults with schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a severely disabling brain disorder. People with schizophrenia often experience hallucinations, delusions, thought disorders, and movement disorders. Physical activity (PA) has been shown not only to increase quality of life, but also to reduce risk factors for several chronic diseases and conditions. The majority of adults, however, do not engage in the recommended amount of PA. Research has shown that people with schizophrenia are even less likely to be regularly physically active. Symptoms of schizophrenia, pharmacological treatments for the disease, and the lifestyle associated with the disease tend to contribute to physical inactivity and the resulting complications. Effective interventions to increase PA have been developed for the general adult population, but very little is known about how to adapt them for use in adults with schizophrenia. The PRIME (Physically Ready for Invigorating Movement Every Day) program is a lifestyle intervention focused on increasing physical activity. This study will evaluate the effectiveness of a modified PRIME program in reducing the risk for morbidity in sedentary adults with schizophrenia.

Participants in this 24-week, single-blind study will be randomly assigned to either the PRIME intervention group or the comparison group, which will involve the Program for Activity, Leisure Skills, and Socialization (PALSS). All participants will attend 90-minute sessions weekly for the first 16 weeks, then biweekly for the remaining 8 weeks. PRIME sessions will focus on learning about PA, setting PA-related goals, and assessing short- and long-term goals. Goals may include early-stage process-oriented goals, such as reading about PA benefits or finding a walking partner. Goals tailored to later stages of change include explicit PA goals, such as increasing frequency, duration, and intensity of PA. Training will also be accomplished online and via printed material. PALSS sessions will focus on motivating participants to engage in leisure and social activity. Sessions will include interactive, structured activity that will be led by a therapist, as well as unstructured leisure activities, such as board games, cards, general socialization, and viewing a travel video. Social and communication skills will not be explicitly taught or practiced. All participants will attend study visits at Months 2, 6, and 8 to assess outcomes. A follow-up visit will be held 2 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Speaks English
* Diagnosis of schizophrenia or schizoaffective disorder
* Currently living in a residential facility
* Currently receiving outpatient care
* Medical clearance
* Willing to sign a release of medical information

Exclusion Criteria:

* Inability to complete assessments
* Medical conditions that may make increasing physical activity unsafe
* Pregnant
* Currently participating in regular moderate to vigorous physical activity (defined as more than 150 minutes per week)

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2006-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Frequency and intensity of PA | Measured at baseline and Months 2, 6, and 8

SECONDARY OUTCOMES:
Quality of life | Measured at baseline and Months 2, 6, and 8
Body mass index (BMI) | Measured at Months 2, 6, and 8
Blood pressure | Measured at baseline and Months 2, 6, and 8

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Lindamer, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States